CLINICAL TRIAL: NCT04916925
Title: Effect of Vitamin D Oral Supplementation in Poly Cystic Ovarian Women Resistant to Clomiphene Citrate
Brief Title: Effect of Vitamin D Oral Supplementation in Poly Csytic Ovarian Women Resistant to Clomiphene Citrate
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: rana alaaeldin aly ibrahim nasr (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, rana alaaeldin aly ibrahim nasr, Clinical gynecology professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCOS resistant to CC & vit D
Record Dates: First submitted 2019-07-21; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Vitamin D Deficiency; Clomiphene Allergy; Polycystic Ovary Syndrome
Keywords: Poly cystic ovary syndrome; Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency; Polycystic Ovary Syndrome | interventions — Vitamin D; Clomiphene

STUDY DESIGN:
Intervention Model Description: a single arm clinical trail
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pcos resistant to cc plus vit d (Experimental): 100 patients who are PCOS and resist CC will receive Vitamin D 10000 IU orally plus 150mg clomid orally for 3 months number and size of growing follicles will be monitored
  Interventions: Drug: Vitamin D; Drug: Clomid

INTERVENTIONS:
Drug: Vitamin D — Adding vitamin D to PCOS patients who are resistant to clomiphene regime for induction will or not improve the Clinical pregnancy rate and will or not increase chances of ovulation and pregnancy.
Drug: Clomid — CLOMID is adrug used for ovulation induction

SUMMARY:
effect of vitamin D oral supplementation in poly csytic ovarian women resistant to clomiphene citrate

DETAILED DESCRIPTION:
Polycystic ovarian syndrome is the most common endocrine disorder . It is associated with chronic anovulation and infertility. The diagnosis is made by clinical and ancillary investigations revealing the presence of irregular menstrual cycles, an ovulation , Hyperandrgenemia , and the presence of polycystic ovaries (ovarian morphology as the presence of 12 or more follicles measuring 2-9 mm in diameter and an increased ovarian volume >10 cm 3) ovulation can be induced with clomiphene citrate (CC), However, ~20%-25% of anovulatory women with PCOS do not respond to CC and are considered to be "clomiphene-resistant( clomiphene citrate resistance means failure to ovulate with 3 months use of clomid at 150 mg/day for 5 days ) Vitamin D may serve as a key in preventing and attenuating the insulin resistance. Vitamin D plays a physiologic role in reproduction including ovarian follicular development and luteinisation, follicle-stimulating hormone sensitivity and progesterone production in human granulosa cells. It also affects glucose homeostasis .

In this trial 100 women with PCO disease that diagnosed by ROTTERDAM CRITERIA (must have any TWO of This findings: Hyperandrogenism, Oligomenorrhea, Polycystic ovaries). Who are taking clomiphene citrate for induction of ovulation and resistant to it, which means failure to ovulate with 3 months of usage of clomid at 150 mg/day for 5 days. They will recieve vitamin D (ossofortin®, Eva Pharma) orally 10000 IU twice weekly for other three months period with clomiphene citrate orally 150 mg/day for 5 days. Number and size of the growing follicles will be monitored before and after taking vitamin D by trans-vaginal ultrasound at day11-14 of the cycle till day 21 to detect effect of vitamin D in ovulation rate.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years 2- Polycystic ovarian syndrome diagnosis made according to ESHRE/ASRM criteria.

  1. Polycystic ovaries (either 12 or more follicles or increased ovarian volume [> 10 cm3
  2. Oligo-ovulation or anovulation
  3. Clinical and/or biochemical signs of hyperandrogenism (Azziz, 2006). 3- PCOS infertile women resistant to CC for 3 cycles. clomiphene citrate resistance means failure to ovulate with 3 months use of clomid at 150 mg/day for 5 days

Exclusion Criteria:

* Causes of infertility other than PCOS.

  1. Male factor.(normal semen analysis)
  2. Other factors e.g. endometriosis
  3. Tubal factor. (normal hysterosalpingography)
  4. Premature ovarian failure: Day 3 FSH > 14 mlu/ml or antimullerian hormone <1 ng/ml.
  5. Normal ultrasound except for criteria of PCO
* Causes of anovulation other than PCOS.
* Patients with hyperprolactinemia
* Patients with thyroid dysfunction.
* Current or in last six months use of vit D treatment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — in child bearing age
Enrollment: 100 (Estimated)
Dates: Start 2021-08-21 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
number of the ovulated follicles | 36 hours of taking HCG injection
  Number of ovulated follicles by trans vaginal ultra sound signs of ovulation

SECONDARY OUTCOMES:
pregancy rate | 2 days after delayed menses
  Pregnancy test positive by quantititave see beta HCG level
Evaluation of the endometrial thickness | 36 hour of taking HCG
  Measure the endometrium thickness by transvaginal ultrasound